CLINICAL TRIAL: NCT00000735
Title: A Clinical Trial To Evaluate the Toxicity and Antiviral Effects of a Range of Doses of Ampligen in p24 Antigen Positive HIV-Infected Patients With AIDS or ARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 054; 11028 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; T-Lymphocytes; Infusions, Intravenous; Immunologic Surveillance; Acquired Immunodeficiency Syndrome; ampligen; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — poly(I).poly(c12,U)

INTERVENTIONS:
Drug: Ampligen

SUMMARY:
To determine the safety of intravenous infusion of ampligen in symptomatic HIV-infected patients at several dose levels, to determine the maximum dose that can be tolerated, and to measure the effects of ampligen on the HIV virus infection, immune function, and clinical condition. Ampligen is a suitable drug for clinical trials against HIV because it has been shown to stimulate the immune system and to inhibit replication of HIV in vitro at doses that can be achieved without noticeable harmful side effects.

DETAILED DESCRIPTION:
Ampligen is a suitable drug for clinical trials against HIV because it has been shown to stimulate the immune system and to inhibit replication of HIV in vitro at doses that can be achieved without noticeable harmful side effects.

Patients entered in the study are given ampligen by intravenous infusion at hemophilia treatment centers once during the first week of the trial and twice a week during the following 12 weeks. The dose each patient receives is determined by the responses of earlier patients. If the status of the HIV infection does not improve after the first 13 weeks, ampligen will be stopped. Each patient maintains a daily diary listing any symptoms or problems that occur such as headache, nausea, or change in appetite. Other anti-HIV drugs cannot be taken during the trial, and aspirin or acetaminophen should not be taken for more than 72 hours at any time during the trial without consulting the research staff. Blood will be drawn at intervals during the 13-week trial and 8-week follow-up and used to determine the effect of ampligen on HIV and the immune system as well as to monitor toxicity and side effects.

ELIGIBILITY:
Inclusion Criteria

Hemophiliacs are included. Patients must have:

* Consistently positive serum HIV p24 antigen (= or > 70 pg/ml) defined by the Abbott HIV antigen test. This demonstration must be seen on two occasions, each separated by at least 72 hours, the last of which must be within 2 weeks of starting therapy.
* Positive HIV antibody test.

Prior Medication:

Allowed:

* Acyclovir for short course (7 days).
* Ketoconazole for short course (7 days).
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Trimethoprim / sulfamethoxazole for PCP prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with AIDS encephalopathy as a sole indicator are excluded.

Patients with AIDS encephalopathy as a sole indicator are excluded.

Prior Medication:

Excluded:

* Other experimental medication.
* Antineoplastic therapy.
* Amphotericin B.
* Ganciclovir.
* Excluded within 14 days of study entry:
* Biologic modifiers.
* Corticosteroids.
* Excluded within 30 days of study entry:
* Other antiretroviral agents.
* Excluded within 60 days of study entry:
* Ribavirin.

Active drug or alcohol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyster ME, Study Chair
Locations (2):
- United States (2):
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania

REFERENCES:
- [Background] Armstrong JA, McMahon D, Huang XL, Pazin GJ, Gupta P, Rinaldo CR Jr, Schoenfeld DA, Gaccione P, Tripoli CA, Bensasi S, et al. A phase I study of ampligen in human immunodeficiency virus-infected subjects. J Infect Dis. 1992 Oct;166(4):717-22. doi: 10.1093/infdis/166.4.717. PMID 1527407